CLINICAL TRIAL: NCT03195322
Title: The Use of Complete AlloDerm® Coverage in Two-stage Tissue Expansion and Implant Placement in the Subcutaneous (Pre-pectoral) Plane: a Prospective Pilot
Brief Title: Pre-pectoral AlloDerm® to Reinforce Tissues in Tissue Expander Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00091477
Record Dates: First submitted 2017-04-18; First posted 2017-06-22 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Quality of Life; Breast Cancer; Breast Prosthesis; Pain
Keywords: Immediate Breast Reconstruction; Pain Control; Post Mastectomy Pain Control; Acellular Dermal Matrix
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Breast Neoplasms; Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pre-pectoral Tissue Expander (Experimental): Pre-pectoral immediate tissue expander breast reconstruction with complete AlloDerm® coverage to reinforce breast tissues.
  Interventions: Procedure: Pre-pectoral Tissue Expander

INTERVENTIONS:
Procedure: Pre-pectoral Tissue Expander — All participants in the study will undergo bilateral mastectomy followed by Immediate, bilateral pre-pectoral tissue expander breast reconstruction with complete AlloDerm® coverage.

SUMMARY:
Primary Objective:

• To describe postoperative static pain scores on the Pain Visual Analog Scale at Day 1 in a population of women undergoing bilateral mastectomy followed by immediate, bilateral pre-pectoral tissue expander breast reconstruction reinforced with AlloDerm® coverage.

Secondary Objectives:

* To describe postoperative static and dynamic pain scores on the Pain Visual Analog Scale and Brief Pain Inventory-Short Form at Day 1-60 after tissue expander placement
* To describe nausea/vomiting, and opioid use at Day 1, 2, 3, 7, 30, and 60 after mastectomy and tissue expander placement.
* To describe short-term changes in Quality of Life scores after mastectomy and tissue expander placement.
* To describe postoperative complication rates at Day 1, 2, 3, 7, 30, and 60 after mastectomy and tissue expander placement.
* To describe nausea/vomiting, and opioid use at Day 1, 2, 3, 7, 30, and 60 after final reconstruction with tissue expander exchange for permanent implant.
* To describe short-term changes in Quality of Life scores after final reconstruction with tissue expander exchange for permanent implant.
* To describe postoperative complication rates at Day 1, 2, 3, 7, 30, and 60 after final reconstruction with tissue expander exchange for permanent implant.
* To describe postoperative rates of breast animation deformity at Day 7, 30, and 60 after final reconstruction with tissue expander exchange for permanent implant.
* To describe average hospital length of stay in patients after final reconstruction with tissue expander exchange for permanent implant.
* To describe the patient's final assessment of pre-pectoral reconstruction from free-form text.

Tertiary Objectives:

• To measure cosmetic result and associated residual pain with Alloderm® reinforcement of breast pocket.

DETAILED DESCRIPTION:
Study participants meeting inclusion criteria will be enrolled prior to surgery. Once the patient has been seen by one of the Institutional Review Board (IRB)-approved study physicians at the initial clinic visit and informed consent has been obtained, pre-study patient-reported outcome (PRO) questionnaires will be distributed and collected by one of the IRB-approved healthcare providers (i.e. medical assistant, nurse, nurse-practitioner, or plastic surgeon). These questionnaires include the Pain Visual Analog Scale, the Patient Pain Assessment Questionnaire which assesses static and dynamic pain as well as nausea and interference with sleep, the Subjective Pain Survey, the preoperative Breast-Q: Reconstruction Module, the SF-36, and the Brief Pain Inventory-Short Form. Participants will then be asked to complete a general patient history form.

Patients will undergo bilateral mastectomy followed by immediate, bilateral pre-pectoral tissue expander breast reconstruction with complete AlloDerm® coverage. Patients who are determined to be poor surgical candidates intra-operatively will be excluded from the study and receive standard of care reconstruction. All patient-specific surgical details will be recorded intra-operatively. See Figure 1 for a schematic of the first stage of reconstruction: bilateral mastectomy and tissue expander placement.

Following the surgery, postoperative pain will be assessed by the Pain Visual Analog Scale (VAS), the Patient Pain Assessment Questionnaire, and the Brief Pain Inventory-Short Form (BPI-SF); pain medication/opioid use and nausea/vomiting will be assessed by the Postoperative nausea and vomiting (PONV) Intensity Scale; and adverse events (AEs)/serious adverse events (SAEs) and the occurrence of complications (seroma, hematoma, cellulitis, and infection requiring expander removal) will be assessed by staff during the hospital stay (Day 1, Day 2, Day 3) and on Day 7 (±2 days) when participants return to clinic for the first follow-up visit after mastectomy and tissue expander placement. At this visit on Day 7, an updated medical history will be completed, pain medication and opioid use will be recorded, and participant complications/AEs/SAEs assessed. In order to minimize missing data, participants will be educated by an IRB-approved member to complete all possible questionnaire items. Furthermore, in order to avoid expectancy-bias, study team members will ensure that patients complete the PRO questionnaires before meeting with study healthcare providers for all postoperative follow-up appointments. Following the completion of all assessments on Day 7, patients will undergo initiation of tissue expander expansion carefully recording the rate and volume of fill.

Longer-term quality-of-life/health outcomes assessments will be performed on postoperative Day 30 (±4 days) and Day 60 (±7 days) after the initiation of tissue expander expansion. During these visits, pain scores (Pain Visual Analog Scale, Patient Pain Assessment Questionnaire, and Brief Pain Inventory-Short Form), pain medication/opioid use, postoperative Breast-Q, and SF-36 questionnaires will be administered. Day 60 follow-up is included as a tertiary endpoint to capture differences in residual pain. Patients will be asked to complete the same questionnaires as at the Day 30 follow-up.

Following final reconstruction with tissue expander exchange for permanent implant, typically three months after mastectomy and tissue expander placement, all PRO questionnaires, postoperative static and dynamic pain, nausea/vomiting/opioid use, short-term changes in Quality of Life, complication rates, average hospital length of stay and residual pain will be assessed. Additionally, on Day 30, and Day 60 after permanent implant placement patients will be photographed comparing the breasts at rest and with pectoralis muscle flexion to assess for breast animation deformity using the Spear 4-point grading system. They will then be imaged using "VECTRA® XT 3D" digital imaging technology ("CANFIELD Scientific", Inc.) on Day 60. Differences in breast volume, surface area, shape, size, contour, and symmetry will be evaluated using the "VECTRA® XT" Analysis Module software. Day 60 follow-up is included as a tertiary endpoint to capture differences in cosmetic result and residual pain after final reconstruction. Patients will be asked to complete the same questionnaires as at the Day 30 follow-up. See Figure 2 for a schematic of the second stage of reconstruction: tissue expander exchange for permanent implant.

*Patients will be called the morning of their Day 7, Day 30, and Day 60 appointments as a reminder. In the event they are unable to attend, every attempt will be made to reschedule within 2, 4, and 7 days, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Be women, aged 18-75 years.
* Choose bilateral mastectomy (therapeutic or prophylactic) followed by immediate, bilateral pre-pectoral tissue expander breast reconstruction with complete AlloDerm® coverage.
* Have no inflammatory breast cancers.
* Be aware of the nature of her malignancy.
* Understand the study purpose, requirements, and risks.
* Be able and willing to give informed consent.

Exclusion Criteria:

* Plan to undergo final reconstruction with autologous material.
* Allergies to gentamicin, cefoxitin, lincomycin, vancomycin, or polymixin (antibiotics used in the pre-treatment of AlloDerm®).
* Active connective tissue disease.
* Current smokers.
* History of, or plan to undergo irradiation of the breasts.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Postoperative Static Pain Score in patients receiving pre-pectoral Tissue Expander placement for Breast Reconstruction using Visual Analog Scale (VAS) | Day 1
  Postoperative static pain scores with standard deviations from VAS will be measured on post-operative (after mastectomy and tissue expander placement) at Day 1

SECONDARY OUTCOMES:
Evaluation of Postoperative Dynamic Pain Score in patients receiving pre-pectoral Tissue Expander placement for Breast Reconstruction using VAS | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60
  Postoperative dynamic pain scores with standard deviations from VAS will be measured on post-operative (after mastectomy and tissue expander placement) Day 1, Day 2, Day 3, and Day 7, before the initiation of tissue expander expansion, and in post-operative Day 30, and Day 60 following initiation of tissue expander expansion.
Evaluation of Postoperative Static Pain Score in patients receiving pre-pectoral Tissue Expander placement for Breast Reconstruction using VAS | Day 2, Day 3, Day 7, Day 30, and Day 60
  Postoperative static pain scores with standard deviations from VAS will be measured on post-operative (after mastectomy and tissue expander placement at Day 2, Day 3, and Day 7, before the initiation of tissue expander expansion, and in post-operative Day 30, and Day 60 following initiation of tissue expander expansion.
Evaluation of Postoperative Static Pain Score in patients receiving pre-pectoral Tissue Expander placement for Breast Reconstruction using "BPI-SF" questionnaire | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60
  postoperative static pain scores with standard deviations from BPI-SF, will be measured on post-operative (after mastectomy and tissue expander placement) Day 1, Day 2, Day 3, and Day 7 before the initiation of tissue expander expansion, and in post-operative Day 30, and Day 60 following initiation of tissue expander expansion.
Level of Postoperative opioid use after Mastectomy and Tissue Expander | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60
  Evaluation of level of opioids (type of opioids and dosage) which the patient required to alleviate the pain related to the insertion and expansion of tissue expander. Relevant information will be assessed by the patients' charts (when inpatient) and by patients' reports to study members (as an outpatient) on Day 1, Day 2, Day 3, Day, 7, Day 30, and Day 60 after mastectomy and tissue expander placement.
Number of participants with postoperative vomiting after Mastectomy and Tissue Expander placement using the PONV Intensity Scale | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60
  Evaluation of number of participants who report postoperative vomiting according to the PONV Intensity Scale at Day 1, Day 2, Day 3, Day, 7, Day 30, and Day 60 after mastectomy and tissue expander placement.
Number of participants with postoperative nausea after Mastectomy and Tissue Expander placement using the PONV Intensity Scale | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60
  Evaluation of number of participants who report postoperative nausea to either according the PONV Intensity Scale at Day 1, Day 2, Day 3, Day, 7, Day 30, and Day 60 after mastectomy and tissue expander placement.
Evaluation of Postoperative Quality of Life scores of patients receiving tissue expander placement by using Breast-Q questionnaire | Day 30
  Postoperative short-term changes in Quality of Life scores by using the Breast-Q questionnaire scores, on Day 30 after mastectomy and tissue expander placement.
Evaluation of Changes in Postoperative Quality of Life scores of patients receiving tissue expander placement by using Breast-Q questionnaire | Baseline and Day 30
  Preoperative and postoperative (Day 30 after mastectomy and tissue expander placement) Quality of Life scores will be assessed by using the Breast-Q questionnaire scores. Changes in Quality of Life Scores will be assessed by subtracting preoperative score from the one recorded postoperative.
Evaluation of Postoperative Quality of Life scores of patients receiving tissue expander placement by using SF-36 questionnaire | Day 7, Day 30
  Postoperative short-term changes in Quality of Life scores by using the SF-36 Health Survey, after mastectomy and tissue expander placement on post-operative Day 7, and Day 30.
Evaluation of Changes in Postoperative Quality of Life scores of patients receiving tissue expander placement by using SF-36 questionnaire | Day 7, Day 30
  Preoperative and postoperative (Day 7, 30 after mastectomy and tissue expander placement) Quality of Life scores will be assessed by using the SF-36 Health Survey. Changes in Quality of Life Scores will be assessed by subtracting preoperative score from the ones recorded postoperative.
Number of participants with any postoperative complication following mastectomy and tissue expander placement based on the Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60
  Postoperative complication rates will be assessed by patients' charts at Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after mastectomy and tissue expander placement. Number and characteristics of complications will be recorded.
Level of Postoperative opioid use after final breast reconstruction | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after final reconstruction
  Evaluation of level of opioids (type of opioids and dosage) which the patient required to alleviate the pain related to final breast reconstruction with permanent implant. Relevant information will be assessed by the patients' charts (when inpatient) and by patients' reports to study members (as an outpatient) on Day 1, Day 2, Day 3, Day, 7, Day 30, and Day 60 after final reconstruction with permanent implant.
Number of participants with postoperative vomiting after final breast reconstruction using the PONV Intensity Scale | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after final reconstruction
  Evaluation of number of participants who report postoperative vomiting according to the PONV Intensity Scale at Day 1, Day 2, Day 3, Day, 7, Day 30, and Day 60 after final breast reconstruction with permanent implant.
Number of participants with postoperative nausea after final breast reconstruction using the PONV Intensity Scale | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after final reconstruction
  Evaluation of number of participants who report postoperative nausea according to the PONV Intensity Scale at Day 1, Day 2, Day 3, Day, 7, Day 30, and Day 60 after final breast reconstruction with permanent implant
Evaluation of Postoperative Quality of Life scores of patients receiving final breast reconstruction with permanent implant by using Breast-Q questionnaire | Day 30, 60
  Postoperative short-term changes in Quality of Life scores by using the Breast-Q questionnaire scores, on Day 30, and Day 60 after final breast reconstruction with permanent implant.
Evaluation of Changes in Postoperative Quality of Life scores of patients receiving final breast reconstruction by using Breast-Q questionnaire | Day 30, 60
  Preoperative, postoperative after mastectomy and tissue expander placement and postoperative after final breast reconstruction Quality of Life scores will be assessed by using the Breast-Q questionnaire scores. Changes in Quality of Life Scores will be assessed by subtracting the most recent score from the previous one, and the most recent from the very first one.
Evaluation of Postoperative Quality of Life scores of patients receiving final breast reconstruction by using SF-36 questionnaire | Day 7, Day 30, Day 60
  Postoperative short-term changes in Quality of Life scores by using the SF-36 Health Survey, after final breast reconstruction at post-operative Day 7, Day 30, and Day 60.
Evaluation of Changes in Postoperative Quality of Life scores of patients receiving final breast reconstruction by using SF-36 questionnaire | Day 7-60
  Preoperative, postoperative after mastectomy and tissue expander placement and postoperative after final breast reconstruction Quality of Life scores will be assessed by using the SF-36 Health Survey. Changes in Quality of Life Scores will be assessed by subtracting the most recent score from the previous one, and the most recent from the very first one.
Number of participants with any postoperative complication following final breast reconstruction based on the Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after final reconstruction
  Postoperative complication rates will be assessed by patients' charts at Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after final breast reconstruction with permanent implant. Number and characteristics of complications will be recorded.
Number of participants with postoperative breast animation deformity assessed by Spear grading system and "VECTRA XT 3D" | Day 7, Day 30, Day 60
  Postoperative rates of breast animation deformity will be assessed at Day 7, Day 30, and Day 60 after final reconstruction with permanent implant, using the Spear 4-point grading system. Participants will then be imaged using VECTRA® XT 3D digital imaging technology ("CANFIELD Scientific, Inc.") on Day 60. Differences in breast volume, surface area, shape, size, contour, and symmetry will be evaluated using the "VECTRA® XT" Analysis Module software
Evaluation of Hospital Length of Stay after final reconstruction in days | Day 1-3
  Hospital Length of Stay in days after final reconstruction with permanent implant will be assessed and recorder by reviewing patients' chart
Evaluation of Postoperative Static Pain Score in patients receiving final Breast Reconstruction using Visual Analog Scale (VAS) | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after final reconstruction
  Postoperative static pain scores with standard deviations from VAS will be measured on post-operative at Day 1, Day 2, Day 3, and Day 7, Day 30, and Day 60 following final breast reconstruction.
Evaluation of Postoperative Dynamic Pain Score in patients receiving final Breast Reconstruction using Visual Analog Scale (VAS) | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after final reconstruction
  Postoperative dynamic pain scores with standard deviations from VAS will be measured on post-operative at Day 1, Day 2, Day3, and Day 7, Day 30, and Day 60 following final breast reconstruction.
Evaluation of Postoperative Static Pain Score in patients receiving final Breast Reconstruction using BPI-SF | Day 1, Day 2, Day 3, Day 7, Day 30, and Day 60 after final reconstruction
  Postoperative static pain scores from BPI-SF will be measured on post-operative at Day 1, Day 2, Day3, and Day 7, Day 30, and Day 60 following final breast reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Gedge D Rosson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
At the moment, there is no plan to share Individual Participant Data (IPD)

REFERENCES:
- [Background] American Cancer Society. Breast Cancer Facts and Figures 2015-2016. http://www.cancer.org. Accessed November 5, 2015.
- [Background] Lucas DJ, Sabino J, Shriver CD, Pawlik TM, Singh DP, Vertrees AE. Doing more: trends in breast cancer surgery, 2005 to 2011. Am Surg. 2015 Jan;81(1):74-80. PMID 25569069
- [Background] Albornoz CR, Bach PB, Mehrara BJ, Disa JJ, Pusic AL, McCarthy CM, Cordeiro PG, Matros E. A paradigm shift in U.S. Breast reconstruction: increasing implant rates. Plast Reconstr Surg. 2013 Jan;131(1):15-23. doi: 10.1097/PRS.0b013e3182729cde. PMID 23271515
- [Background] Edsander-Nord A, Brandberg Y, Wickman M. Quality of life, patients' satisfaction, and aesthetic outcome after pedicled or free TRAM flap breast surgery. Plast Reconstr Surg. 2001 Apr 15;107(5):1142-53; discussion 1154-5. doi: 10.1097/00006534-200104150-00007. PMID 11373553
- [Background] Girotto JA, Schreiber J, Nahabedian MY. Breast reconstruction in the elderly: preserving excellent quality of life. Ann Plast Surg. 2003 Jun;50(6):572-8. doi: 10.1097/01.SAP.0000069064.68579.19. PMID 12783001
- [Background] Harless C, Jacobson SR. Current strategies with 2-staged prosthetic breast reconstruction. Gland Surg. 2015 Jun;4(3):204-11. doi: 10.3978/j.issn.2227-684X.2015.04.22. PMID 26161305
- [Background] Susarla SM, Ganske I, Helliwell L, Morris D, Eriksson E, Chun YS. Comparison of clinical outcomes and patient satisfaction in immediate single-stage versus two-stage implant-based breast reconstruction. Plast Reconstr Surg. 2015 Jan;135(1):1e-8e. doi: 10.1097/PRS.0000000000000803. PMID 25539329
- [Background] Sbitany H, Sandeen SN, Amalfi AN, Davenport MS, Langstein HN. Acellular dermis-assisted prosthetic breast reconstruction versus complete submuscular coverage: a head-to-head comparison of outcomes. Plast Reconstr Surg. 2009 Dec;124(6):1735-1740. doi: 10.1097/PRS.0b013e3181bf803d. PMID 19952627
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841
- [Background] Spear SL, Schwartz J, Dayan JH, Clemens MW. Outcome assessment of breast distortion following submuscular breast augmentation. Aesthetic Plast Surg. 2009 Jan;33(1):44-8. doi: 10.1007/s00266-008-9275-y. Epub 2008 Dec 4. PMID 19052809
- [Background] Vardanian AJ, Clayton JL, Roostaeian J, Shirvanian V, Da Lio A, Lipa JE, Crisera C, Festekjian JH. Comparison of implant-based immediate breast reconstruction with and without acellular dermal matrix. Plast Reconstr Surg. 2011 Nov;128(5):403e-410e. doi: 10.1097/PRS.0b013e31822b6637. PMID 22030500
- [Background] Reitsamer R, Peintinger F. Prepectoral implant placement and complete coverage with porcine acellular dermal matrix: a new technique for direct-to-implant breast reconstruction after nipple-sparing mastectomy. J Plast Reconstr Aesthet Surg. 2015 Feb;68(2):162-7. doi: 10.1016/j.bjps.2014.10.012. Epub 2014 Oct 16. PMID 25455288
- [Background] Lee KT, Mun GH. Updated Evidence of Acellular Dermal Matrix Use for Implant-Based Breast Reconstruction: A Meta-analysis. Ann Surg Oncol. 2016 Feb;23(2):600-10. doi: 10.1245/s10434-015-4873-9. Epub 2015 Oct 5. PMID 26438439
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Kim MS, Sbalchiero JC, Reece GP, Miller MJ, Beahm EK, Markey MK. Assessment of breast aesthetics. Plast Reconstr Surg. 2008 Apr;121(4):186e-194e. doi: 10.1097/01.prs.0000304593.74672.b8. PMID 18349598
- [Background] LifeCell Corporation, USA. AlloDerm® Regenerative Tissue Matrix: Instructions for Use. (http://www.lifecell.com/fileadmin/media/files/downloads/Alloderm_IFU_D.pdf)
- [Background] Memorial Sloan-Kettering Cancer Center. QScore Scoring Software [Internet]. US; 2012 [cited 2016 Apr 19]. Available from: https://webcore.mskcc.org/breastq/scoring.html
- [Background] Optum, Inc. SF-36v2 Health Survey [Internet]. US; 2016 [cited 2016 Apr 19]. Available from: https://www.optum.com/optum-outcomes/what-we-do/health-surveys/sf-36v2-health-survey.html
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Cleeland C. Brief Pain Inventory User Guide. Houston: University of Texas M. D. Anderson Cancer Center; 2009.
- [Background] Mathias SD, Crosby RD, Qian Y, Jiang Q, Dansey R, Chung K. Estimating minimally important differences for the worst pain rating of the Brief Pain Inventory-Short Form. J Support Oncol. 2011 Mar-Apr;9(2):72-8. doi: 10.1016/j.suponc.2010.12.004. PMID 21542414